CLINICAL TRIAL: NCT03296540
Title: COMPARison of Pre-hospital CRUSHed vs. Uncrushed Prasugrel Tablets in Patients With STEMI Undergoing Primary Percutaneous Coronary Interventions
Brief Title: CRUSHed vs. Uncrushed Prasugrel in STEMI Patients Undergoing PCI
Acronym: CompareCrush
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Collaborators: MicroPort Orthopedics Inc. (Industry); Daiichi Sankyo (Industry); Research Maatschap Cardiologen Rotterdam Zuid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-40
Record Dates: First submitted 2017-09-06; First posted 2017-09-28 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Cardiovascular Diseases
Keywords: STEMI
MeSH Terms: conditions — Cardiovascular Diseases; ST Elevation Myocardial Infarction | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Intervention Model Description: Crushed versus uncrushed tablets Prasugrel loading dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uncrushed (Active Comparator): 6 Integral tablets Prasugrel as loading dose
  Interventions: Drug: Prasugrel (Integral tablets)
- Crushed (Experimental): 6 Crushed tablets Prasugrel as loading dose
  Interventions: Drug: Prasugrel (Crushed tablets)

INTERVENTIONS:
Drug: Prasugrel (Crushed tablets) — loading dose of 6 crushed tablets 10mg Prasugrel
  Other Names: 6 Crushed tablets of Prasugrel 10mg
  Arms: Crushed
Drug: Prasugrel (Integral tablets) — loading dose of 6 integral tablets of 10mg Prasugrel
  Other Names: 6 Integral tablets of Prasugrel 10mg
  Arms: Uncrushed

SUMMARY:
The studys evaluates the effect of prehospital administration of crushed tablets of Prasugrel loading dose (in addition to ASA and standard care) versus uncrushed tablets of Prasugrel loading dose on efficacy and safety as well as pharmacodynamics as measured by platelet reactivity using VerifyNow.

DETAILED DESCRIPTION:
The study is a two-centre, randomized, 1:1 trial comparing prehospital prasugrel initiation therapy between crushed vs. uncrushed prasugrel tablets on efficacy and safety as well as pharmacodynamics in STEMI patients.

Patients with STEMI planned for primary PCI will be screened and, if inclusion criteria are met, included at first medical contact (paramedics). After enrolment, patients will be randomly assigned (1:1) to receive 60mg prasugrel loading dose by ingesting integral or crushed tablets.

The follow-up duration is 12 months, i.e. clinical outcomes will be analysed in-hospital, at 30 days, and 12 months

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients with STEMI planned for primary PCI:

* Deferred written informed consent within 4 hours after prasugrel loading dose
* Adult men and women aged at least 18 years
* Symptoms of acute MI of more than 30 min but less than 6 hours
* New persistent ST-segment elevation ≥ 1 mm in two or more contiguous ECG leads

Exclusion Criteria:

* Contraindication to prasugrel (e.g., hypersensitivity, active bleeding, history of previous intracranial bleed, history of any CVA including TIA, moderate to severe hepatic impairment, GI bleed within the past 6 months, major surgery within past 4 weeks)
* Patient who has received loading dose of clopidogrel or ticagrelor for the index event or are on chronic treatment of ticagrelor, or prasugrel. However, patients on maintenance dose clopidogrel for at least 7 days are included in the study (see appendix A).
* Oral anticoagulation therapy that cannot be stopped (i.e. patients requiring chronic therapy)
* Planned fibrinolytic treatment
* Patient requiring dialysis
* Known, clinically important thrombocytopenia
* Known clinically important anaemia
* Known pregnancy or lactation
* Need for a concomitant systemic therapy with strong inhibitors or strong inducers of CYP3A
* Condition which may either put the patient at risk or influence the result of the study (e.g., cardiogenic shock with severe hemodynamic instability, active cancer, risk for non-compliance, risk for being lost to follow up)
* Patient unable to swallow oral medication (i.e. intubated patients)
* Patient who have not received prasugrel loading dose in the ambulance
* Patient who vomited after randomization / receiving the loading dose prasugrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 729 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Co-primary endpoint is the percentage of patients reaching TIMI flow grade 3 of MI culprit vessel at initial angiography or a ≥70% ST-segment resolution directly post-PCI | directly post PCI
  To assess the efficacy of crushed vs. integral tablets of prasugrel loading dose treatment by comparing the percentage of patients reaching the co-primary endpoint of TIMI flow grade 3 of MI culprit vessel at initial angiography or a ≥70% ST-segment elevation resolution directly post-PCI.

SECONDARY OUTCOMES:
Composite of death, MI, stroke, urgent revascularization and acute stent thrombosis in hospital, at 30 days and 12 months | upto 72 hours after randomisation, at 30 days and 12 months.
  Percentage of patients in the following: composite of death, MI, stroke, urgent revascularization and acute stent thrombosis during inhospital stay, 30 days and 12 months of study
Composite of death, MI, urgent revascularization during inhospital, at 30 days and 12 months of study | 30 days and 12 months
  Percentage of patients in the following: composite of death, MI, or urgent revascularization during inhospital, 30 days and 12 months of study
Individual endpoints during inhospital, at 30 days and 12 months of study | upto 72 hours after randomisation, at 30 days and 12 months.
  Percentage of patients presenting with any of the individual endpoints during inhospital, 30 days and 12 months of study
Thrombotic bail-out with GPIIb/IIIa inhibitors at initial PCI | directly post PCI
  Percentage of patients receiving thrombotic bail-out with GPIIb/IIIa inhibitors at initial PCI
Complete (≥ 70%) ST-segment elevation resolution pre-PCI and 60 min post-PCI | pre-PCI and 60 min post-PCI
  Complete (≥ 70%) ST-segment elevation resolution pre-PCI and 60 min post-PCI
Corrected TIMI frame count (cTFC) at angiography, pre and post PCI. | pre PCI, directly post PCI
  Corrected TIMI frame count (cTFC) at angiography, pre and post PCI
TIMI myocardial perfusion grade (TMPG) at angiography, pre and post PCI. | pre PCI, directly post PCI
  TIMI myocardial perfusion grade (TMPG) at angiography, pre and post PCI.
Time-relationship (from symptom onset to 1st dose intake) on each co-primary | directly post-PCI
  Time from symptom onset to 1st dose intake correlated to TIMI flow grade 3 of MI culprit vessel at initial angiography and on ≥70% ST-segment elevation resolution directly post-PCI
Time-relationship (from 1st dose intake to ECG/ angiography) on each co-primary | directly post-PCI
  Time from first dose intake to ECG correlated to ≥70% ST-segment elevation resolution directly post-PCI and time from randomization to initial angiography correlated to TIMI flow grade 3 of MI culprit vessel
TIMI flow grade 3 at end of procedure. | directly post PCI
  TIMI flow grade 3 at end of procedure.
Myocardial Blush at the start and end of the procedure | pre PCI, directly post PCI
  Myocardial Blush at the start and end of the procedure
Maximum CK, and CK-MB levels | upto 72 hours after randomisation
  Maximum CK, and CK-MB levels
Level of platelet inhibition at first medical contact, beginning and end of PCI procedure, as well as at 4 hours after prasugrel administration | at time of prasugrel administration, pre PCI, directly post PCI, 4 hours after prasugrel administration
  Level of platelet inhibition at first medical contact, beginning and end of PCI procedure, as well as at 4 hours after prasugrel administration
Platelet reactivity, at each time point as well as over time | at time of prasugrel administration, pre PCI, directly post PCI, 4 hours after prasugrel administration
  PRU measurements at first medical contact, beginning and end of PCI, as well as 4hours after drug administration
Rates of HPR | upto 72 hours after randomisation
  Percentage of patients with PRU values over HPR threshold
Exploratory analyses within each group to evaluate any differences in PD among patients receiving morphine | upto 72 hours after randomisation
  PD of each group among patients stratified for morphine treatment

CONTACTS AND LOCATIONS:
Overall Officials: George Vlachojannis, MD, PhD, Principal Investigator — Maasstadziekenhuis; Pieter C Smits, MD, PhD, Study Director — Maasstadziekenhuis; Nicolas van Mieghem, MD, PhD, Study Chair — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam
  - Maasstadziekenhuis, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vlachojannis GJ, Wilschut JM, Vogel RF, Lemmert ME, Delewi R, Diletti R, van der Waarden NWPL, Nuis RJ, Paradies V, Alexopoulos D, Zijlstra F, Montalescot G, Angiolillo DJ, Krucoff MW, Van Mieghem NM, Smits PC. Effect of Prehospital Crushed Prasugrel Tablets in Patients With ST-Segment-Elevation Myocardial Infarction Planned for Primary Percutaneous Coronary Intervention: The Randomized COMPARE CRUSH Trial. Circulation. 2020 Dec 15;142(24):2316-2328. doi: 10.1161/CIRCULATIONAHA.120.051532. Epub 2020 Oct 14. PMID 33315489
- [Derived] Vlachojannis GJ, Vogel RF, Wilschut JM, Lemmert ME, Delewi R, Diletti R, van Vliet R, van der Waarden N, Nuis RJ, Paradies V, Alexopoulos D, Zijlstra F, Montalescot G, Angiolillo DJ, Krucoff MW, Van Mieghem NM, Smits PC. COMPARison of pre-hospital CRUSHed vs. uncrushed Prasugrel tablets in patients with STEMI undergoing primary percutaneous coronary interventions: Rationale and design of the COMPARE CRUSH trial. Am Heart J. 2020 Jun;224:10-16. doi: 10.1016/j.ahj.2020.03.005. Epub 2020 Mar 11. PMID 32272255